CLINICAL TRIAL: NCT04543916
Title: A Phase 1/2 Study of Venetoclax and Irinotecan in Relapsed/Refractory Small Cell Lung Cancer
Brief Title: Venetoclax and Irinotecan in Relapsed/Refractory SCLC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: AbbVie decided to stop trial involving Venetoclax for safety measures needed
Sponsor: Virginia Commonwealth University (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17-13842; HM20019851 (Other: Virginia Commonwealth University Massey Cancer Center)
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Relapsed Small Cell Lung Cancer; Refractory Small Cell Lung Carcinoma
Keywords: Relapsed SCLC; Refractory SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — venetoclax; Irinotecan

STUDY DESIGN:
Intervention Model Description: Dose escalation will proceed within each cohort. Phase II is the expansion cohort at the recommended phase 2 dose found in phase 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Level 1 (Experimental): Venetoclax 50mg by mouth once daily and Irinotecan 60 mg/m2 intravenously (IV) on days 1, 8, and 15
  Interventions: Drug: Venetoclax 50 MG; Drug: Irinotecan 60 mg/m2
- Dose Level 2 (Experimental): Venetoclax 100mg by mouth once daily and Irinotecan 60 mg/m2 intravenously (IV) on days 1, 8, and 15
  Interventions: Drug: Venetoclax 100 MG; Drug: Irinotecan 60 mg/m2
- Dose Level 3 (Experimental): Venetoclax 200mg by mouth once daily and Irinotecan 60 mg/m2 intravenously (IV) on days 1, 8, and 15
  Interventions: Drug: Venetoclax 200 MG; Drug: Irinotecan 60 mg/m2
- Dose Level 4 (Experimental): Venetoclax 400mg by mouth once daily and Irinotecan 60 mg/m2 intravenously (IV) on days 1, 8, and 15
  Interventions: Drug: Venetoclax 400; Drug: Irinotecan 60 mg/m2
- Dose Level 5 (Experimental): Venetoclax 600mg by mouth once daily and Irinotecan 60 mg/m2 intravenously (IV) on days 1, 8, and 15
  Interventions: Drug: Venetoclax 600; Drug: Irinotecan 60 mg/m2
- Phase 2 Expansion Cohort (Experimental): Venetoclax recommended phase 2 dose (RP2D) by mouth once daily and Irinotecan 60 mg/m2 intravenously (IV) on days 1, 8, and 15
  Interventions: Drug: Irinotecan 60 mg/m2; Drug: Venetoclax (RP2D)

INTERVENTIONS:
Drug: Venetoclax 50 MG — Escalating doses to determine recommended phase 2 dose (RP2D)
  Arms: Dose Level 1
Drug: Venetoclax 100 MG — Escalating doses to determine recommended phase 2 dose (RP2D)
  Arms: Dose Level 2
Drug: Venetoclax 200 MG — Escalating doses to determine recommended phase 2 dose (RP2D)
  Arms: Dose Level 3
Drug: Venetoclax 400 — Escalating doses to determine recommended phase 2 dose (RP2D)
  Arms: Dose Level 4
Drug: Venetoclax 600 — Escalating doses to determine recommended phase 2 dose (RP2D)
  Arms: Dose Level 5
Drug: Irinotecan 60 mg/m2 — Intravenously (IV), days 1, 8, and 15
Drug: Venetoclax (RP2D) — orally, once per day
  Arms: Phase 2 Expansion Cohort

SUMMARY:
This study is a single-arm, open-label, multicenter phase 1/2 trial designed to establish the recommended phase 2 dose (RP2D) of daily oral venetoclax when given in combination with irinotecan in patients with relapsed or refractory small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
Irinotecan will be given at 60 mg/m2 on days 1, 8, and 15 of each 28-day cycle. A 3+3 dose escalation design will be followed until the maximum tolerated dose (MTD) of venetoclax has been determined. Once the MTD is established, a RP2D that is the same as or less than the MTD will be determined. If no RP2D can be determined, the study will close to accrual. The RP2D will be used in an expansion cohort based on a Simon's two-stage minimax design to evaluate efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of SCLC
* Disease progression or recurrence during or after platinum-based therapy, unless platinum-based therapy was contraindicated
* Phase 1: Measurable or evaluable disease according to RECIST v1.1
* Phase 2: Measurable disease according to RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Age ≥ 18 years
* Adequate bone marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 8.0 g/dL
* Adequate renal function as defined below:
* Serum creatinine ≤ upper limit of normal (ULN) for the lab or a calculated creatinine clearance ≥ 40 mL/min
* Adequate hepatic function as defined below:

  * Total bilirubin ≤ 1.5 x ULN for the laboratory
  * Aspartate aminotransferase (AST) ≤ 2.5 x ULN for the laboratory
  * Alanine aminotransferase (ALT) ≤ 2.5 x ULN for the laboratory
* Persons with known HIV seropositivity are eligible if they meet the following criteria:

  * CD4 count ≥ 200/mm3
  * Undetectable HIV viral load on standard PCR-based test
  * On a stable regimen of highly active anti-retroviral therapy (HAART) that does not include protocol contraindicated agents
  * No ongoing requirement for concurrent antibiotics or antifungal agents for the prevention of HIV-associated opportunistic infections
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Ongoing requirement for any non-study anticancer therapy
* Ongoing or planned treatment with any of the following:

  * Greater than 10 mg prednisone daily or equivalent
  * Immunosuppressive agents
  * Strong or moderate CYP3A inhibitor or inducer, or a narrow-therapeutic sensitive substrate
  * P-gp inhibitor or narrow-therapeutic sensitive P-gp substrate If any of these agents have been used, patients must be off them for ≥ 1 week before initiation of study treatment.
* Any investigational agent within 21 days prior to the first dose of the investigational drugs
* Has consumed grapefruit, grapefruit products, Seville oranges, or starfruit within 3 days before initiation of study treatment.
* Phase 2 portion only: Previous systemic anticancer therapy other than platinum-based therapy
* Known leptomeningeal metastases
* Known untreated brain metastases
* Hypersensitivity to irinotecan, venetoclax, or their excipients
* Diarrhea ≥ grade 1
* Ongoing need for antidiarrheal agents
* Active uncontrolled infection, ongoing or within 2 weeks before initiating treatment
* Known homozygosity for the UGT1A1*28 allele Note: Study-specific UGT1A1 testing is not required
* Inability to swallow oral medications and/or malabsorption
* Pregnancy or breastfeeding
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Determine the recommended phase 2 dose (RP2D) of venetoclax with irinotecan in patients with relapsed or refractory SCLC | 90 Days
  Recommended phase 2 dose (RP2D) of venetoclax in combination with irinotecan that is less than or equal to the maximum tolerated dose (MTD). A 3+3 dose escalation design will be followed until the maximum tolerated dose (MTD) of venetoclax has been determined. Patients assigned to a dose level of venetoclax greater than 50 mg will undergo a ramp-up phase during the first week of irinotecan
Phase 2: Evaluate the efficacy of venetoclax with irinotecan in patients with relapsed or refractory SCLC | 180 Days
  The RP2D will be used in an expansion cohort based on a Simon's two-stage minimax design to evaluate efficacy.

SECONDARY OUTCOMES:
Assess the frequency of adverse events (AEs) | 120 Days
  Assess adverse events (AEs) characterized and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE V 5.0) to determine safety and toxicity of the combination of venetoclax and irinotecan.
Evaluate the antitumor effects of venetoclax and irinotecan in combination. | 180 Days
  Evaluate the anti tumor effects of tumor response based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
Observe survival in relapsed or refractory SCLC patients receiving venetoclax in combination with irinotecan | 180 Days
  Progression-free survival and overall survival of patients with relapsed or refractory SCLC receiving venetoclax in combination with irinotecan

CONTACTS AND LOCATIONS:
Overall Officials: Sosipatros Boikos, MD, Principal Investigator — Massey Cancer Center